CLINICAL TRIAL: NCT07306871
Title: Subendometrial Injection Versus Intrauterine Infusion of Platelet Rich Plasma for Women With Recurrent Implantation Failure A Prospective Randomized Controlled Study
Brief Title: Subendometrial Injection Versus Intrauterine Infusion of Platelet Rich Plasma for Women With Recurrent Implantation Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed mouner saber, Assistant lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1551991
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-05

CONDITIONS: Recurrent Implantation Faliure; Infertility
Keywords: Platelet Rich Plasma; Recurrent impantation failure
MeSH Terms: conditions — Infertility | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subendometrial PRP group (Active Comparator): 4 ml PRP will be injected in this group into the sub endometrial space(1-2 ml)below endometrium at multiple sites trans vaginally & through the cervix after insertion of a cuscow speculum via ovum pick up needle under ultrasound guidance in the luteal phase of previous cycle of FET.
  Interventions: Biological: Platelet rich plasma
- Intrauterine infusion group (Active Comparator): Intrauterine infusion of 4 ml PRP will be done during FET cycle when endometrium reaches 7 mm.
  Interventions: Biological: Platelet rich plasma
- Control group (Active Comparator): will undergo standard FET with no intervention only hormonal preparation .
  Interventions: Other: No intervention /standard care

INTERVENTIONS:
Biological: Platelet rich plasma — Autologous platelet-rich plasma prepared from peripheral blood and administered either by subendometrial injection or intrauterine infusion prior to embryo transfer.
  Arms: Intrauterine infusion group; Subendometrial PRP group
Other: No intervention /standard care — Participants will receive standard IVF/ICSI care without platelet-rich plasma administration.
  Arms: Control group

SUMMARY:
Aim of this study is to compare the effectiveness of subendometrial PRP injection & intrauterine PRP infusion in women with recurrent implantation failure in comparison with a control group .

DETAILED DESCRIPTION:
This prospective randomized cotrolled study will be conducted in Private IVF centers in Minia governorate from January 2024 till December 2025,after being approved by the local Ethical committee of the department & written informed consent will be obtained from participants .

All patients will be counselled regarding inclusion in this study ,a written informed consent will be taken from each patient prior to participation in this study.

Recruited patients will be randomly allocated into 3 groups using opaque sealed closed envelops .

Sample size:

Based on previous studies & by using the sample size calculation of GPower software version 3.1.9.6 (Franz Faul, Kiel university, Germany), and setting β at 95% and α at 0.05. This makes sample size of 47 per each group. This figure will be rounded 25. Assuming a drop- out rate of 12%, this will make sample size 60 per each group.

(Group1)-(subendometrial PRP group )SE-PRP(n=60): 4 ml PRP will be injected in this group into the sub endometrial space(1-2 ml)below endometrium at multiple sites trans vaginally & through the cervix after insertion of a cuscow speculum via ovum pick up needle under ultrasound guidance in the luteal phase of previous cycle of FET.

(Group 2)-(intrauterine PRP group )IU-PRP(n=60) Intrauterine infusion of 4 ml PRP will be done during FET cycle when endometrium reaches 7 mm.

(GROUP 3)The control group(n=60) will undergo standard FET with no intervention only hormonal preparation .

Endometrial preparation :

For all groups The Endometrium will be prepared by combined estrogen and progesterone protocol as approved by IVF centeres. Estradiol valerate will be started on day 2/3 of FET cycle at dose of 6mg with measurement of endometrial thickness on the 10 th day of the cycle and every 48 houres & once endometrium is >7mm progesterone vaginal pessary 400 mg twice daily will be offered for luteal support for 3-5 days then embryos of the same number & same quality (grade A top quality embryos ) will be transferred in all patients . Estradiol and progesterone will be continued after the transfer till the 12th week of gestational age if pregnancy occurred.

PRP preparation :

PRP will be prepared from autologous blood using a modified two step centrifuge process. , 8.5 ml of peripheral venous blood will be drawn in the syringe that contained 1.5 ml of Acid Citrate A Anticoagulan solution (ACD-A) and centrifuged immediately at 1600 g for 10 min. The blood will be divided into three layers: red blood cells at the bottom, cellular plasma in the supernatant and a buffy coat layer between them. The plasma layer and buffy coat will be collected to another tube and centrifuged again at 3500 g for 5 min to obtain 1.5 ml PRP with 4-5 times more concentrated .

ELIGIBILITY:
Inclusion Criteria:

* Age 18 -40 years .
* BMI<30 Kg/m2.
* An IVF procedure resulting in at least one top quality embryo .
* At least one cancelation history of embryo transfer due to thin endometrium (failure of achieving 7 mm endometrial thickness in the cycle) in frozen embryo transfer (FET) cycles after receiving standard hormone therapy.
* Women had a history of failure to achieve pregnancy after two or more embryo transfers with high-quality embryos.

Exclusion Criteria:

* women with other factors that may affect implantation success are excluded: ;

  * BMI >30 kg/m2.
  * Untreated uterine abnormalities.
  * untreated hydrosalpinges.
  * Thrombophilia.
  * uncontrolled endocrinopathy
  * severe male factor infertility.
  * difficult embryo transfer.
  * only poor quality embryos available .
  * couple with chromosomal abnormalities
  * Hematological disorders (blood cancer ,thrombocytopenia )
  * Hormonal disorders (DM,thyroid disorders )
  * Immunological disorders (anti phospholipid syndrome).
  * renal failure
  * Genetic ,chromosomal abnormalities

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Implantation rate | 5 weeks after embryo transfer
  the ratio of gestational sacs to the number of embryos transferred .

SECONDARY OUTCOMES:
Chemical pregnancy rate | 14 days after embryo transfer
  serum B-hCG 50 IU/L after 14 days from embryo transfer.
Clinical pregnancy rate | 5 weeks after embryo transfer
  the presence of a gestational sac with heart beat identified by ultrasound 5 weeks after the embryo transfer.

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code